CLINICAL TRIAL: NCT06287866
Title: Pinch Grafting Versus Second Intention Wound Healing for Mohs Micrographic Surgery Defects on the Scalp
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2099470
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Scarring
Keywords: Pinch graft
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Two blinded observers will record their scores independently using the POSAS instrument.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Second Intention Wound Healing (No Intervention)
- Pinch Grafting (Experimental)
  Interventions: Procedure: Pinch Graft

INTERVENTIONS:
Procedure: Pinch Graft — In the pinch graft technique, the investigators will numb and then shave off a thin piece of skin and place it in the wound bed.
  Arms: Pinch Grafting

SUMMARY:
Oftentimes, following surgery on the scalp, wounds are left to heal by themselves. This is called "second intention." Open wounds left to heal on the scalp often take 8 weeks or more to completely heal. The investigators are investigating how second intention closure compares to another established reconstruction technique, called "pinch graft." In the pinch graft technique, a dermatological surgeon numbs and then shaves off a thin piece of skin (usually from the groin area) and places it in the wound bed it (also known as "grafting"), to encourage growth of new healthy skin. This study will compare time-to-healing in the second intention method versus the pinch graft method.

DETAILED DESCRIPTION:
Pinch graft methodology was first developed in 1976 as a treatment to accelerate healing of lower leg ulcerations, particularly venous or gravitational ulcerations (1, 2). It was later adapted as a tool to hasten healing in surgical wounds, such as surgical closure of diabetic foot wounds (3). It has also been used in the healing of patients with wounds related to dystrophic epidermolysis bullosa (4). More recently, pinch grafts have been investigated as a reconstruction option for Mohs micrographic surgery defects (5). In this study, patients with below the knee Mohs surgical defects were randomized to receive either PG reconstruction or SIH reconstruction. Patients with PG reconstruction healed 20 days sooner (i.e., faster time to reepithelialization) than those who underwent SIH. Complication rates, including infection and reported pain, were also lower in the PG cohort compared to the SIH cohort. SIH is often recommended as a reconstruction technique for surgical wounds without adjacent skin laxity to support primary closure, such as the anterior lower extremity and scalp. There is no study to date examining the use of pinch grafts in scalp wounds. In our study, the investigators explore whether PG is a viable and useful reconstruction method for wounds on the scalp that otherwise would be left to close via SIH. Specifically, in our study, the investigators examine the comparative time to healing and complication rates between PG and SIH in Mohs surgical defects of the scalp.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure on the scalp with predicted second intention closure
* Willing to return for follow up visit
* Active user of MyChart
* Willing to send weekly messages until wound is healed

Exclusion Criteria:

* Incarceration
* Under 18 years of age
* Pregnant women
* Unable to understand written and oral English
* Scalp wounds with planned primary repair reconstruction
* Surgical defects with bone exposure
* No MyChart access or use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to re-epithelialization | 1-8 weeks
  Participants will submit weekly photos to blinded reviewers to assess for re-epithelization.

SECONDARY OUTCOMES:
Observer Scar Assessment as measured by Patient Observer Scar Assessment Score (POSAS) | 3 months
  The primary endpoint will be the score of two blinded reviewers independently using the POSAS assessment. The observer scale of the POSAS consists of six items (vascularity, pigmentation, thickness, relief, pliability, and surface area). All items are scored on a scale ranging from 1 ("like normal skin") to 10 ("worst scar imaginable"). The sum of the six items results in a total score of the POSAS observer scale. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10. All parameters should preferably be compared to normal skin on a comparable anatomic location.
Patient Scar Assessment as measured by Patient Observer Scar Assessment Score (POSAS) | 3 months
  This is the patient portion of the POSAS assessment, which will be independently recorded. The patient scale of the POSAS consists of six items (pain, itch, thickness, color, stiffness, and irregularity). All items are scored on a scale ranging from 1 ("as normal skin") to 10 ("yes, very different"). The sum of the six items results in a total score of the POSAS patient scale. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, MD, Principal Investigator — University of California, Davis - Dermatology
Locations (1):
- University of California, Davis - Dermatology Department, Sacramento, California, United States

REFERENCES:
- [Background] Burns DA, Sarkany I. Management of stasis ulcers by pinch graft. Br J Dermatol. 1976 Jul;95 Suppl 14:82. doi: 10.1111/j.1365-2133.1976.tb07931.x. No abstract available. PMID 776204
- [Background] Millard LG, Roberts MM, Gatecliffe M. Chronic leg ulcers treated by the pinch graft method. Br J Dermatol. 1977 Sep;97(3):289-95. doi: 10.1111/j.1365-2133.1977.tb15185.x. PMID 336073
- [Background] Ramanujam CL, Zgonis T. Pinch graft harvesting technique for surgical closure of the diabetic foot. Clin Podiatr Med Surg. 2012 Oct;29(4):585-8. doi: 10.1016/j.cpm.2012.07.004. Epub 2012 Aug 30. PMID 23044064
- [Background] Claude O, Binder JP, Bustamante K, Blanchet-Bardon C, Andrivon F, Revol M, Servant JM. [Role of cutaneous pinch grafts in the healing of patients with dystrophic epidermolysis bullosa wounds: report of four cases]. Ann Chir Plast Esthet. 2005 Jun;50(3):189-96. doi: 10.1016/j.anplas.2004.11.010. Epub 2004 Dec 18. French. PMID 15963838
- [Background] Willenbrink TJ, Brodland DG. Pinch Grafts Versus Second Intention Wound Healing for Mohs Micrographic Surgery Defects Below the Knee: A Prospective Randomized Trial. Dermatol Surg. 2024 Nov 1;50(11):1010-1016. doi: 10.1097/DSS.0000000000004272. Epub 2024 Aug 1. PMID 39088685
- [Background] Joo J, Custis T, Armstrong AW, King TH, Omlin K, Kappel ST, Eisen DB. Purse-string suture vs second intention healing: results of a randomized, blind clinical trial. JAMA Dermatol. 2015 Mar;151(3):265-70. doi: 10.1001/jamadermatol.2014.2313. PMID 25372450